CLINICAL TRIAL: NCT01095289
Title: Electromyographic Activity of Masseter Muscle During Deglutition in Total Laryngectomized Subjects
Status: Completed | Type: Observational
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Hilton Justino da Silva, Federal University of Pernambuco
Other Study IDs: emgca-01
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-01

CONDITIONS: Head and Neck Cancer
Keywords: electromyography; laryngeal neoplasms; masticatory muscles
MeSH Terms: conditions — Head and Neck Neoplasms; Laryngeal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Total Laryngectomized

SUMMARY:
The objective of this study is to evaluate the electromyographic activity of masseter muscle during deglutition in laryngectomized subjects.

ELIGIBILITY:
Inclusion Criteria:

* laryngectomy

Exclusion Criteria:

* neurological diseases
* no oral feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 16 subjects underwent total laryngectomy
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leandro Pernambuco, Graduated, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Cancer Hospital of Pernambuco, Recife, Pernambuco, Brazil

REFERENCES:
- [Derived] Pernambuco Lde A, Silva HJ, Nascimento GK, Silva EG, Balata PM, Santos Vda S, Leao JC. Electrical activity of the masseter during swallowing after total laryngectomy. Braz J Otorhinolaryngol. 2011 Sep-Oct;77(5):645-50. doi: 10.1590/s1808-86942011000500018. PMID 22030975